CLINICAL TRIAL: NCT03548025
Title: Safety and Efficacy of the BTL-FR2000 Device for the Treatment of Facial Wrinkles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-786-001
Record Dates: First submitted 2018-03-28; First posted 2018-06-06 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Treated group of subjects, serves as its own control
  Interventions: Device: BTL-703 (Treatment group)

INTERVENTIONS:
Device: BTL-703 (Treatment group) — Treatment with BTL-FR2000 Device

SUMMARY:
The study will evaluate safety and effectivity of the BTL-FR2000 device for the treatment of facial wrinkles.

DETAILED DESCRIPTION:
Subjects will be photographed at the baseline visit. After the treatment phase, subjects will be invited for two follow-up visits - 3 and 6 months after the last therapy. They will be again photographed.

Three blinded evaluators will be scoring the full face photos according to the Fitzpatrick Wrinkle Severity Scale. The improvement of the scores will be evaluated. Every subject will serve as its own control.

In addition, the occurence of an AE during the whole study, as well as the therapy discomfort during the treatment phase, will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 years
* Voluntarily signed informed consent form

Exclusion Criteria:

* Bacterial or viral infection, acute inflammations
* Impaired immune system
* Isotretinoin in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and chemotherapy
* Poor healing and unhealed wounds in the treatment area
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any kind of cancer
* Active collagen diseases
* Cardiovascular diseases (such as cardiac and vascular diseases, peripheral arterial disease, thrombophlebitis, thrombosis, etc.)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Children under age of 21
* Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks
* Patients with allergy to anesthetics should not be treated under anesthesia
* Botox®/collagen/fat injections or other injected bio-material in the treated area within three months prior to treatment
* Use of non-steroidal anti-inflammatory drugs one week before and after each treatment session
* Treating over tattoo or permanent makeup

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of facial wrinkles evaluated through the change in the value of the validated scale | 10 months
  Three blinded evaluators will be evaluating the full-face photographs taken at the baseline, last therapy visit and both follow-up visits. They will be evaluating it using the validated Fitzpatrick Wrinkle Severity Scale. According to that scale, subjects are divided in three categories (I, II, III) corresponding to mild, moderate, and severe wrinkling, and degree of elastosis. In addition, a score of 1 to 9 (a linear sliding scale to represent increasing severity of wrinkling) will be given.
  The change in score (value) from the scale before and after the treatment will be calculated.

SECONDARY OUTCOMES:
Safety - Occurence of AE | 10 months
  The occurence of serious AE during the whole study will be followed.
Safety - Therapy comfort | 4 months
  The discomfort during the therapy will be evaluated immediately after every therapy, using the Discomfort Questionnaire. Subjects will be asked to evaluate the agreement with the statement concerning the conformity of the study treatment. Subjects will be evaluating the agreement by choosing an answer on a scale between 1 (Strongly disagree) and 5 (Strongly agree). Based on a given answers, the therapy comfort will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Aesthe Clinic, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No